CLINICAL TRIAL: NCT00471757
Title: Etiology of Community Acquired Pneumonia
Acronym: CAP
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: PRO07040291
Record Dates: First submitted 2007-05-09; First posted 2007-05-10 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Streptococcus Pneumonia; Haemophilus Influencae; Mycoplasma Pneumonia; Chlamydia Pneumonia
Keywords: pnuemonia; influenca
MeSH Terms: conditions — Pneumonia; Pneumonia, Mycoplasma; Psittacosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The proposed study aims to provide current information, etiology and outcome of community-acquired pneumonia (CAP), risk factors for for CAP in isolates of Streptococcus pneumoniae and Haemophilus influencae, Mycoplasma pneumoniae, chlamydia pneumoniae and Legionella. Risk factors, including patient demographics, comorbid illnesses, setting of presentation, causative organisms, antibiotic history, and resistance profiles will be assessed and outcome will be recorded.

DETAILED DESCRIPTION:
The following information will be collected: age, sex, occupation, hospital location at the time of positive culture (ER, medical ward, ICU etc), date of positive culture, prior hospitalization, receipt of outpatient dialysis, home care or other regular medical care (eg, outpatient chemotherapy), presence of invasive devices, receipt of antibiotics, including their type and whether they were adequate for the resistance profile of the organism, prior positive microbiologic cultures, time and location of positive cultures, underlying diseases and severity of illness, co-morbid illnesses, presence of urinary or intravascular devices, recent immunomodulative therapies or radiation therapy, physical exam findings, laboratory and radiographical data, antimicrobial usage within 30 days of onset of the infection, microbiological data and resistance patterns, choice of antibiotics once organism identified, bacteriological outcomes, laboratory results, demographic information, medications, clinical outcome,gender, height, weight, ethnicity, and past medical history. We will collect information retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* All patients with Streptococcus pneumoniae, Haemophilus influencae, Mycoplasma pneumoniae, chlamydia pneumoniae and Legionella species infections during the time period the study will be reviewed. A community-associated pneumonia isolate will be defined as one which was recovered from a clinical culture from a patient at UPMC who had no established risk factors for infection with an antibiotic resistant organism. Established risk factors are defined as: Isolation of the organism two or more days after admission for hospitalization OR history of hospitalization, surgery, dialysis, or residence in a long-term care facility within one year before the culture date OR The presence of an indwelling catheter or percutaneous medical device (eg, tracheostomy tube, gastrostomy tube, or Foley catheter) at the time of the culture OR Previous isolation of an antibiotic resistant organism.

Exclusion Criteria:

* Does not meet entry criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: streptococcus pneumoniae positive
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L Paterson, MD, Principal Investigator — University of Pittsburgh/University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
not sharing